CLINICAL TRIAL: NCT00608231
Title: Dexmedetomidine Effects on Microelectrode Recording in Deep Brain Stimulation
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Intraoperative recording could not be maintained for required period
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Joseph Neimat, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 070666
Record Dates: First submitted 2008-01-07; First posted 2008-02-06 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson's Disease; Essential Tremor; Dystonia
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- PD-STN (Experimental): Parkinson's Disease -- STN target
  Interventions: Drug: Dexmedetomidine Hydrochloride Infusion
- PD - GPi (Experimental): Parkinson's Disease -- GPi target
  Interventions: Drug: Dexmedetomidine Hydrochloride Infusion
- ET - VIM (Experimental): Essential Tremor -- VIM target
  Interventions: Drug: Dexmedetomidine Hydrochloride Infusion
- Dystonia - GPi (Experimental): Dystonia -- GPi target
  Interventions: Drug: Dexmedetomidine Hydrochloride Infusion
- PD - STN Control (Placebo Comparator): Parkinson's Disease -- STN target
  Interventions: Drug: Normal Saline
- PD - GPi Control (Placebo Comparator): Parkinson's Disease -- GPi target
  Interventions: Drug: Normal Saline
- ET - VIM Control (Placebo Comparator): Essential Tremor -- VIM target
  Interventions: Drug: Normal Saline
- Dystonia - GPi Control (Placebo Comparator): Dystonia -- GPi target
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride Infusion — Dexmedetomidine Hydrochloride Infusion(0.5-1.0 mg/kg)intravenous over 10 minutes with dose adjustment for goal Richmond Agitation and Sedation Scale of -1 During deep brain stimulator implantation surgery
  Other Names: Precedex
  Arms: Dystonia - GPi; ET - VIM; PD - GPi; PD-STN
Drug: Normal Saline — Normal Saline intravenous over 10 minutes during deep brain stimulator implantation surgery
  Other Names: Placebo control
  Arms: Dystonia - GPi Control; ET - VIM Control; PD - GPi Control; PD - STN Control

SUMMARY:
To test the hypothesis that sedation induced by Dexmedetomidine at levels appropriate for awake, DBS surgery has no significant effect on electrophysiological parameters of DBS micro-electrode recordings

DETAILED DESCRIPTION:
Deep brain stimulator (DBS) implants are used in the treatment of medically refractory movement disorders such as Parkinson's disease, essential tremor and dystonia. Because of the uniqueness of each individual brain, the surgery to implant a DBS electrode requires detailed anatomic and physiological information for each patient. The anatomic data is obtained before surgery via a Magnetic Resonance Imaging (MRI) scan of the patient's brain. Physiological data is obtained during the operation via micro-electrode recording of the patient's brain and neurological examination of the patient. Therefore, DBS surgery can be uncomfortable to patients, as it can be very time consuming and requires the patient to be awake and attentive.

The specific aims of this project are:

1. To test the hypothesis that sedation induced by Dexmedetomidine at levels appropriate for awake, DBS surgery has no significant effect on electrophysiological parameters of DBS micro-electrode recordings.
2. To test the hypothesis that sedation induced by Dexmedetomidine at levels appropriate for awake, DBS surgery have no significant effects on neurological findings and/or patient cooperation during neurological examination.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has agreed to undergo DBS implantation.

Exclusion Criteria:

* Patients who fail recommendation for DBS surgery discussed in Vanderbilt University Movement Disorder Clinical Conference.
* Patients not consented for DBS surgery.
* Patients or legal guardians not able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Micro-electrode Recordings | Intra-operative

SECONDARY OUTCOMES:
Neurological Exam Findings | Intra-operative

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Neimat, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States